CLINICAL TRIAL: NCT01347398
Title: Validity of a Supersimplified Device for Diagnosis of Patients With Suspected Obstructive Sleep Apnoea-hypopnoea (OSAH).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Hospital Txagorritxu (Joaquín Duran Cantolla), Basque Health Service
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ApneaLink
Record Dates: First submitted 2011-04-18; First posted 2011-05-04 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep apnoea; Diagnosis; Blood pressure; Body mass index; Breath analysis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MicroMESAM (Experimental): Sleep study made by MicroMESAM system
  Interventions: Procedure: MicroMESAM system
- PSG (Active Comparator): Sleep study made by PSG (polysomnography)
  Interventions: Procedure: PSG

INTERVENTIONS:
Procedure: PSG — Sleep study made by PSG (polysomnography)
  Arms: PSG
Procedure: MicroMESAM system — Sleep study made by MicroMESAM system
  Arms: MicroMESAM

SUMMARY:
The diagnosis of OSASH requires expensive sleep tests that generate long waiting lists, so we need simplified and rapid diagnostic tools. The ApneaLinkTM, is a device that allows the assessment of respiratory events by measuring the flow ventilation with a nasal cannula connected to a pressure transducer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 to 75 years of both sexes.
2. clinical suspicion of OSAH defined as subjects with breathing pauses during sleep and / or asphyxiated sounds, with or without excessive daytime sleepiness as measured by the Epworth scale and who have asked for a sleep test to rule out OSAH.
3. Informed consent signed by the patient.

Exclusion Criteria:

1. Place of residence more than 100 km from the hospital.
2. inability to perform psychophysical study at home.
3. cardio-vascular disease, cerebro-vascular or respiratory or acute severe unstable as to preclude the proper conduct of studies at home and / or PSG in the laboratory.
4. Patients with chronic insomnia or recognize sleep less than six hours.
5. Patients with depression (both point 4 and 5 are the potential causes of false negatives in a PR for lack of sufficient sleep time).
6. nasal obstruction complete or nearly complete, which prevents obtaining a quality signal with MicroMESAM

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients correctly diagnosed by MicroMESAM (APNEA-LINK) | 3 months

REFERENCES:
- [Derived] Masa JF, Duran-Cantolla J, Capote F, Cabello M, Abad J, Garcia-Rio F, Ferrer A, Fortuna AM, Gonzalez-Mangado N, de la Pena M, Aizpuru F, Barbe F, Montserrat JM; Spanish Sleep Network. Efficacy of home single-channel nasal pressure for recommending continuous positive airway pressure treatment in sleep apnea. Sleep. 2015 Jan 1;38(1):13-21. doi: 10.5665/sleep.4316. PMID 25325508
- [Derived] Masa JF, Duran-Cantolla J, Capote F, Cabello M, Abad J, Garcia-Rio F, Ferrer A, Mayos M, Gonzalez-Mangado N, de la Pena M, Aizpuru F, Barbe F, Montserrat JM; Spanish Sleep Network; Larrateguy LD, de Castro JR, Garcia-Ledesma E, Utrabo I, Corral J, Martinez-Null C, Egea C, Cancelo L, Garcia-Diaz E, Carmona-Bernal C, Sanchez-Armengol A, Fortuna AM, Miralda RM, Troncoso MF, Monica G, Martinez-Martinez M, Cantalejo O, Pierola J, Vigil L, Embid C, Del Mar Centelles M, Prieto TR, Rojo B, Vanesa L. Effectiveness of home single-channel nasal pressure for sleep apnea diagnosis. Sleep. 2014 Dec 1;37(12):1953-61. doi: 10.5665/sleep.4248. PMID 25325484